CLINICAL TRIAL: NCT05566028
Title: A Randomized, Double-blind, Multi-center, Therapeutic Confirmatory, Phase 3 Trial to Evaluate the Efficacy and Safety of D150, D745 and D759 Combination Therapy in Pateints with Type 2 Diabetes Inadequately Controlled with D150 Plus D759
Brief Title: The Efficacy and Safety of D745 Added to D150 Plus D759 Therapy in Patients with Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A127_02DM2210
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Expermental group 1 (Experimental): Pateints assigned to this group are treated with D150, D759 and D745 formulation I
  Interventions: Drug: D745 formulation I
- Experimental group 2 (Experimental): Pateints assigned to this group are treated with D150, D759 and D745 formulation II
  Interventions: Drug: D745 formulation II
- Placebo group (Placebo Comparator): Pateints assigned to this group are treated with D150, D759 and D745 placebo
  Interventions: Drug: D745 Placebo

INTERVENTIONS:
Drug: D745 formulation I — QD for 24 weeks or 52 weeks(if extension study) with D150 and D759
  Arms: Expermental group 1
Drug: D745 formulation II — QD for 24 weeks or 52 weeks(if extension study) with D150 and D759
  Arms: Experimental group 2
Drug: D745 Placebo — QD for 24 weeks or 52 weeks(if extension study) with D150 and D759
  Arms: Placebo group

SUMMARY:
The purpose of this study is to prove that the group treated with D745 in combination added that the reduction of HbA1c superior to placebo treated group added in combination.

DETAILED DESCRIPTION:
The aim of this phase 3 study is to evaluate the efficacy and safety of additional combined D745 administration for 24 weeks in patient with type 2 diabetes who are no adequately controlled for blood glucose by the combination of D150 and D759

ELIGIBILITY:
Inclusion Criteria:

* between 19 years and 85 years old(male or female)
* Type 2 diabetes mellitus
* BMI between 18.5kg/m2 and 40kg/m2
* Agreement with written informed consent

Exclusion Criteria:

* Type 1 diabetes mellitus or secondary diabetes mellitus
* Patients with complications of severe diabetes such as proliferative diabetic retinopathy
* Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Patients with abnormal laboratory test results according to the protocol
* Continuous or non continuous treatment insulin within 12 weeks prior to screening
* Chronic oral or non oral corticosteroids treatment within 4 weeks prior to screening

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | Baseline, 24 week

SECONDARY OUTCOMES:
Change from baseline in HbA1c | Baseline, 12 week
Change from baseline in Fasting plasma glucose | Baseline, 12 week, 24 week

CONTACTS AND LOCATIONS:
Overall Officials: Youngmin Cho, M.D, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No